CLINICAL TRIAL: NCT00175110
Title: The Effect of Hibiscus Sabdariffa L. Tisane on Blood Pressure in Prehypertensive and Mildly Hypertensive Men and Women
Brief Title: The Effect of Hibiscus Sabdariffa L. Tea on Blood Pressure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Celestial Seasonings (Industry); Tufts Medical Center (Other)
Responsible Party: Jeffrey B. Blumberg, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PV3727
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: pre-hypertension; mild hypertension
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — Phytotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: herbal therapy/botanical therapy (Hibiscus sabdariffa)

SUMMARY:
The goal of this study is to find out whether the plant compounds present in Hibiscus sabdariffa, a plant commonly used in herbal tea blends and other beverages, will have a beneficial effect on blood pressure in people with mildly elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure 120-150 mm Hg
* Diastolic blood pressure 95 mm Hg or less
* Body mass index (BMI) 18.5-34.9 kg/m2

Exclusion Criteria:

* Smoking
* Use of medications that influence blood pressure
* Cardiovascular disease
* Chronic kidney disease
* Diabetes
* Regular use of vitamin C supplements (min 500 mg/day) within prior 30 days
* Regular strenuous aerobic activity greater than 30 min/day
* Excessive intake of caffeine or alcohol
* Pregnancy within last 6 months or during study period
* Abnormal complete blood count (CBC), urinalysis or electrocardiogram (EKG)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Blumberg, Ph.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] McKay DL, Chen CY, Saltzman E, Blumberg JB. Hibiscus sabdariffa L. tea (tisane) lowers blood pressure in prehypertensive and mildly hypertensive adults. J Nutr. 2010 Feb;140(2):298-303. doi: 10.3945/jn.109.115097. Epub 2009 Dec 16. PMID 20018807